CLINICAL TRIAL: NCT06279065
Title: Investigation of the Influence of the Human Microbiome on the Pathogenesis and Recurrence Probability in Giant Cell Arteritis
Brief Title: Investigation of the Influence of the Human Microbiome on Giant Cell Arteritis
Acronym: GCA-Biom
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, Head of the rheumatology department, University Hospital Bonn, University of Bonn
Other Study IDs: 373/23-EP
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Giant Cell Arteritis
Keywords: microbiome
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Blood, oral Lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA Patients: Primary diagnosis of giant cell arteritis
  Interventions: Diagnostic Test: Analysis of blood and microbiome samples (stool, oral lavage)
- Control: Control group without rheumatologic disease
  Interventions: Diagnostic Test: Analysis of blood and microbiome samples (stool, oral lavage)

INTERVENTIONS:
Diagnostic Test: Analysis of blood and microbiome samples (stool, oral lavage) — Analysis of blood and microbiome samples (stool, oral lavage) especially composition of the gut microbiome and potential interaction with immune cells

SUMMARY:
The longitudinal observational study aims to assess the impact of the microbiome especially the gut-microbiome in the emergence and course of giant cell arteritis (abbr. GCA) patients. At diagnosis and 6 month follow up we will analyze the oral, blood and gut microbiome from GCA patients and healthy controls. Thereby identified potential candidate biota will be further analyzed for possible interactions and influence on the immune system.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Giant cell arteritis (only in one arm)

Exclusion Criteria:

* chronic infection (viral, fungi, bacteria) including human immunodeficiency viruses, Hepatitis B/C
* acute infection with usage of antibiotics less then 90 days before screening
* major gastro-intestinal surgery <5 years from screening
* gastro-intestinal bleeding <90 days before screening
* inflammatory bowel disease (confirmed bioptically)
* bulimia or anorexia nervosa
* adipositas (body mass index ≥ 40)
* intake of high dosage of probiotics (>10^9 colony forming units per day) <90 days before screening
* not controlled Diabetes mellitus
* Malignancy within one year (except for squamous skin - and basal skin carcinoma without metastasis, cervix carcinoma with curative surgery, Cutaneous T-cell lymphoma)
* known abuse of alcohol oder drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: no specific requirements, usually over 50 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Significant differences in the composition of the microbiome | At Baseline and 6 month follow up

SECONDARY OUTCOMES:
Influence of the microbiome on therapy response e.g. increased probability of recurrence with accumulation of specific microbiome species | At Baseline and 2 year follow up
potential association of microbiome composition with application of immune modulating drugs | At Baseline and 6 month follow up

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Clinic of Internal Medicine III, Department of Oncology, Haematology, Rheumatology and Clinical Immunology, University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Bonn

IPD SHARING:
Plan to Share IPD: No